CLINICAL TRIAL: NCT02624726
Title: A Open Label, Non Randomized, Phase Two Trial in Metastatic Colorectal Cancer (mCRC) With the Combination of m FOLFIRI Plus Aflibercept as First Line Treatment: MINOAS Trial
Brief Title: Trial in Metastatic Colorectal Cancer With FOLFIRI Plus Aflibercept as First Line Treatment
Acronym: MINOAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/14.01
Record Dates: First submitted 2015-11-24; First posted 2015-12-08 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: 1st line; FOLFIRI; Aflibercept; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI/Aflibercept (Experimental): 5 Fluorouracil/Leucovorin/Irinotecan/Aflibercept
  Interventions: Drug: 5 Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Aflibercept

INTERVENTIONS:
Drug: 5 Fluorouracil — 5 Fluorouracil: 400mg/m2, bolus infusion in <5min followed by 5 Fluorouracil: 2400mg/m2, i.v in 46 hours continuous infusion (cycle repeated every two weeks)
  Other Names: 5 Fluorouracil (5-FU)
Drug: Leucovorin — Leucovorin: 400mg/m2, i.v in 2 hours infusion (cycle repeated every two weeks)
  Other Names: Leucovorin (LV)
Drug: Irinotecan — Irinotecan: 180mg/m2, i.v in 90min infusion (cycle repeated every two weeks)
  Other Names: Irinotecan (CPT-11)
Drug: Aflibercept — Aflibercept: 4mg/kg i.v in 1 hour infusion (cycle repeated every two weeks)
  Other Names: Zaltrap

SUMMARY:
Investigators propose to study the combination of m FOLFIRI plus Aflibercept in a Phase II trial of patients with metastatic colorectal cancer. The promising results of aflibercept derived from preclinical studies and from clinical trials conducted in patients with refractory of recurrent to oxaliplatin-based 1st line treatment in patients with mCRC open the field to explore such therapeutic approaches in the 1st line setting in combination with the FOLFIRI regimen.

DETAILED DESCRIPTION:
Colorectal cancer accounts for 8% of all malignant tumors in adults and is considered as a major cause of cancer morbidity and mortality worldwide. Although curative surgical resection is possible in 70-80% of patients at diagnosis, almost half of them will develop local or/and metastatic recurrence and will die of the disease with the liver been the most common site of metastatic spread from CRC.

Combinations of infusional administrated 5-fluorouracil/Leucovorin with irinotecan or oxaliplatin are accepted as the mainstay of first-line treatment and have increase the median overall survival of patients with advanced CRC from 12 months to about 21-22 months. In addition, resection for colorectal metastases (mainly in the liver), has become the standard of care, for patients with limited metastatic disease confounded to the liver and currently remains the only potentially curative therapy Aflibercept, also known as vascular endothelial growth factor (VEGF) Trap, is an angiogenesis inhibitor with a unique mechanism of action. Aflibercept is a recombinant fusion protein that consists of portions of human VEGFR1 and VEGFR2 extracellular domains fused to the Fc portion of human immunoglobulin G1. This fusion protein binds all forms of Vascular Endothelial Growth Factor-A, as well as VEGF-B and placental growth factor, additional angiogenic growth factors that appear to play a role in tumor angiogenesis and inflammation. Aflibercept has been shown to bind VEGF-A, VEGF-B, and placental growth factor (PlGF) with higher affinity than their native receptors. In vitro and in vivo studies have shown that aflibercept can inhibit new vessel growth and tumor vascularization in tumor models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented adenocarcinomas of colon or rectum with unresectable metastatic disease.
* No prior treatment for metastatic disease
* Metastatic liver disease assessable with diffusion-weighted Magnetic Resonance Imaging (MRI)
* No previous treatment with bevacizumab or Cetuximab or Panitumumab.
* Patients may have receive fluoropyrimidines with or without oxaliplatin as adjuvant treatment, if they have progressed > 12 months after the end of the last cycle of the adjuvant treatment
* Performance Status (ECOG) 0-2
* Life expectancy ≥ 3 months.
* Effective contraception for both male and female subjects if the risk of conception exists.
* Adequate laboratory parameters: Absolute neutrophils count ≥ 1.5 x 109 /L, Platelets ≥ 100 x 109 /L, Leucocytes > 3,000/mm; Hemoglobin> 10.5g/dl, creatinine clearance ≥ 60 ml/min, Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour, Magnesium ≥ lower limit of normal, Calcium ≥ lower limit of normal, total Bilirubin ≤ 1.5 times the upper limit of normal; aspartate and alanine aminotransferase ≤ 3 times of the upper normal limit in absence of liver metastases, or ≤5x Upper Normal Limits (UNL) in presence of liver metastases, alkaline phosphatases < 5x UNL
* All patients will have to sign written informed consent in order to participate in the study.
* Female patients must commit to using reliable and appropriate methods of contraception until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial

Exclusion Criteria:

* Known hypersensitivity reaction to the component of the treatment.
* Inability to underwent a diffusion-weighted MR Imaging at baseline and in predefined time points
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* History or evidence upon physical examination of Central Nervous System (CNS) metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy),
* Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
* Treatment with any other investigational medicinal product within 28 days prior to study entry.
* Other serious and uncontrolled non-malignant disease
* Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy.
* Gilbert's syndrome
* Intolerance to atropine sulfate or loperamide
* Known dihydropyrimidine dehydrogenase deficiency
* Treatment with CYP3A4 inducers unless discontinued > 7 days prior to randomization
* Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis
* Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
* INR in absence of anticoagulation therapy > 1.25 or poorly controlled anti-coagulation therapy on coumadin or heparin compounds (INR >3.0)
* History of myocardial infarction and/or stroke within 6 months prior to randomization, New York Heart Association (NYHA) class III and IV congestive heart failure
* History of life threatening (grade 4) venous thromboembolic events (including pulmonary embolism) within 6 months prior to registration,
* Bowel obstruction
* Legal incapacity or limited legal capacity.
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent.
* A second primary tumour other than non-melanoma skin cancer or in situ cervical cancer.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on chest CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Disease evaluation at Week 8

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Overall Survival | 1 year
Toxicity profile (CTCAE v4.0) | Every 2 weeks up to 100 weeks
  From date of randomization until the date of last follow up or death from any cause, assessed up to 100 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — Hellenic Oncology Research Group; Athanasios Kotsakis, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (10):
- Greece (10):
  - University Hospital of Heraklion Crete, Heraklion, Crete
  - 251 Air Forces Military Hospital of Athens, Athens
  - Anicancer Hospital of Athens "Agios Savvas", Athens
  - Anticanscer Hospital of Athens "Agios Savvas", Athens
  - Athens Hospital "Mitera" Hygia Polis, Athens
  - General Hospital of Athens "Aretaieio", Athens
  - General Hospital of Athens "Sotiria", Athens
  - IASO General Hospital, Athens
  - University Hospital of Patras-Rio, Rio
  - Thessaloniki Bioclinic, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Matikas A, Souglakos J, Katsaounis P, Kotsakis A, Kouroupakis P, Pantazopoulos N, Kentepozidis N, Nikolaidi A, Messaritakis I, Tzovara I, Hatzidaki D, Prinarakis E, Georgoulias V. MINOAS: A Single-arm Translational Phase II Trial of FOLFIRI Plus Aflibercept as First-line Therapy in Unresectable, Metastatic Colorectal Cancer. Target Oncol. 2019 Jun;14(3):285-293. doi: 10.1007/s11523-019-00647-3. PMID 31203498